CLINICAL TRIAL: NCT02716376
Title: Treatment and Prevention of Middle Ear Morbidity in Head and Neck Cancer Patients Following Radiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Jakob Gerlach Christensen, Resident, Zealand University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SJ-435
Record Dates: First submitted 2016-03-03; First posted 2016-03-23 (Estimated); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Otitis Media With Effusion; Chronic Otitis Media; Hearing Loss
Keywords: Head and neck neoplasms; Radiotherapy; Otitis media
MeSH Terms: conditions — Otitis Media with Effusion; Hearing Loss; Head and Neck Neoplasms; Otitis Media

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Otovent® (Experimental): Otovent® is a special designed balloon that is blown up through the nose, also referred to as auto-inflation of the eustachian tube. The patients use the Otovent® 5 times a day.
  Interventions: Device: Otovent®
- No treatment (No Intervention): Observation: No treatment.

INTERVENTIONS:
Device: Otovent® — Otovent® is a special designed balloon that is blown up through the nose, also referred to as auto-inflation of the eustachian tube. The patients use the Otovent® 5 times a day.
  Other Names: Auto-inflation device
  Arms: Otovent®

SUMMARY:
To investigate the incidence of tuba dysfunction (TD) and middle ear (ME) morbidity after radiotherapy (RT) to the Head & Neck and test the effect of auto-inflation of the Eustachian tube (ET) on middle ear effusion with a special designed balloon (Otovent®) and thereby better hearing and ear related quality of life after cancer treatment.

DETAILED DESCRIPTION:
Middle ear complications and TD are common following RT to the Head & Neck, where the radiation field involves the ET and ME. These are due to mucositis and swelling in the surrounding pharyngeal tissue and on the long-term fibrosis. The ET is a small channel from the middle ear to the upper part of the pharynx. It is normally closed but briefly opens while swallowing or yawning. The ME pressure then equalizes and optimize sound conduction to the inner ear. If the function of the ET is impaired it can lead to negative pressure and effusion. This causes pain, tinnitus, otitis media with effusion (OME), chronic otitis media (COM) and hearing loss. Last can be none reversible. Almost everyone experience middle ear morbidity short after RT, but on the long-term up to 20 % have chronic otitis media and TD with significant hearing impairment and the need for hearing aid. Conventional treatment with insertion of ventilation tubes in to the tympanic membrane is not recommended for radiation-induced ME problems.

Methods and materials: The investigators will by randomized controlled trials examine the effect of auto-inflation of the ET on ME morbidity with a custom-made balloon called Otovent®. Examination of the ear is conducted by otoscopy, pure tone and impedance audiometry and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Head and neck cancer patients in Zealand region, Capital region and North Jutland region.
* Only patients who received or is going to receive radiotherapy or chemoradiotherapy as curative intended treatment.
* The irradiated volume involve the nasopharynx.

Exclusion Criteria:

* Patients with documented history of otitis media with effusion or chronic otitis media that is not related to the cancer diagnosis.
* Performance status > 3.
* Surgery in the middle ear, Eustachian tube and surrounding tissue area. (Biopsies during diagnosis is accepted).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Incidence of otitis media with effusion (OME) | 6 months
  Impedance audiometry: A tympanometer I used to measure compliance of the tympanic membrane. Results are presented in a type A, B, or C-curve, with pressure in dekaPascal at the x-axis and compliance in decibel (db) at the y-axis. Type B curve indicates otitis media with effusion.
  B-curve indicate middle ear effusion (OME).

SECONDARY OUTCOMES:
Perforation of the tympanic membrane. | 6 months
  Otoscopy is used to visualize dry perforations of the tympanic membrane.
Chronic suppurative otitis media. | 6 months
  Otoscopy is used to visualize recurrent ear discharges or otorrhoea through a tympanic perforation for more than two weeks.
Hearing loss | 6 months
  Pure tone audiometry: Patient's hearing loss range in decibels (dB HL) presented in an audiogram.
Quality of life after treatment of head and neck cancer. | 6 months
  European Organization for Research and Treatment of Cancer Quality of Life and Head and Neck Module (EORTC-H&N35) questionnaire. Patient related outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Gerlach Christensen, Principal Investigator — Køge University Hospital

IPD SHARING:
Plan to Share IPD: No